CLINICAL TRIAL: NCT01223287
Title: Physiologic Definition of Bronchopulmonary Dysplasia
Acronym: PhysiologicDef
Status: Completed | Type: Observational
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: NICHD-NRN-0032; U10HD027904 (NIH); U10HD021364 (NIH); M01RR000080 (NIH); U10HD027853 (NIH); M01RR008084 (NIH); U10HD040492 (NIH); M01RR000030 (NIH); U10HD027851 (NIH); M01RR000039 (NIH); UL1RR025008 (NIH); U10HD027856 (NIH); M01RR000750 (NIH); UL1RR025761 (NIH); U10HD027880 (NIH); M01RR000070 (NIH); UL1RR025744 (NIH); U10HD053119 (NIH); M01RR000054 (NIH); U10HD034216 (NIH); M01RR000032 (NIH); U10HD040461 (NIH); U10HD053109 (NIH); M01RR000059 (NIH); UL1RR024979 (NIH); U10HD021397 (NIH); M01RR016587 (NIH); U10HD053089 (NIH); M01RR000997 (NIH); U10HD040521 (NIH); M01RR000044 (NIH); UL1RR024160 (NIH); U10HD053124 (NIH); M01RR000064 (NIH); UL1RR025764 (NIH); U10HD040689 (NIH); M01RR000633 (NIH); U10HD021373 (NIH); U10HD040498 (NIH); M01RR007122 (NIH); U10HD021385 (NIH); U10HD027871 (NIH); UL1RR024139 (NIH)
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Bronchopulmonary Dysplasia (BPD)
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Very Low Birth Weight (VLBW); Prematurity; Mechanical ventilation; Chronic Lung Disease (CLD)
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study was conducted to design and test a physiologic definition for bronchopulmonary dysplasia at 36 weeks of life. Infants were studied in a supine position with the pulse oximeter in position with good signal prior to collecting baseline data. Feedings and medications were given 30 minutes before the evaluation. Baseline data was collected on infant's current oxygen. Then, the infants were weaned to room air for 30 minutes. If saturations remain ≥90%, the infant was considered to have passed the oxygen reduction challenge (to NOT have BPD). The infant should then be placed back in his/her baseline oxygen. If the infant has saturations <90% for 5 continuous minutes or <80% for 15 seconds, the infant should be immediately placed back in his/her baseline oxygen, and the infant was considered to have NOT passed the challenge (to have BPD).

DETAILED DESCRIPTION:
One of the confounders to any study that looks at bronchopulmonary dysplasia (BPD) is the lack of a precise definition. Most neonates with BPD do not undergo lung biopsy or any physiologic test; thus, their pulmonary disease is defined clinically, on the basis of the sustained need for supplemental oxygen at 36 weeks postmenstrual age. The validity of this definition is supported by evidence that oxygen dependence at 36 weeks is predictive of long-term impairment in pulmonary function. An inherent limitation of defining BPD by the need for supplemental oxygen is that the need for oxygen is determined by individual physicians, rather than on the basis of a physiologic assessment. Published literature cites acceptable saturation ranges from 88-98%.

This observational study was conducted to design and test a physiologic definition for bronchopulmonary dysplasia at 36 weeks of life.

Infants were studied in a supine position with the pulse oximeter in position with good signal prior to collecting baseline data. Feedings and medications were given 30 minutes before the evaluation. Baseline data was collected on infant's current oxygen. Then, the infants were weaned to room air for 30 minutes. If saturations remain ≥90%, the infant was considered to have passed the oxygen reduction challenge (to NOT have BPD). The infant should then be placed back in his/her baseline oxygen. If the infant has saturations <90% for 5 continuous minutes or <80% for 15 seconds, the infant should be immediately placed back in his/her baseline oxygen, and the infant was considered to have NOT passed the challenge (to have BPD).

ELIGIBILITY:
Inclusion Criteria:

* Infant with birthweight 401-1500 grams
* Alive at 36+1 week corrected age
* On supplemental oxygen as follows:
* A. Infants receiving oxygen by hood at rest:
* A1. Oxygen by hood <27% with majority* of saturations ≥ 90% in prior 24 hours.
* A2. Oxygen by hood 27-30% with majority* of saturations ≥ 96% in prior 24 hours
* B. Infants receiving oxygen by nasal cannula at restΔ:
* B1. Oxygen by nasal cannula <27% EFFECTIVE** oxygen and majority* of saturations ≥90% in prior 24 hours.
* B2. Oxygen by nasal cannula 27-30% EFFECTIVE** oxygen and majority* saturations ≥96% on prior 24 hours.
* C. Infants receiving room air by nasal cannula at ANY liter per minute (lpm) flow.

Exclusion Criteria:

* Need for mechanical ventilation or continuous positive airway pressure (CPAP)
* Oxygen by hood >30%
* Oxygen by nasal cannula >30% effective oxygen

Ages: 36 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants on mechanical ventilation at 36 weeks of life.
Sampling Method: Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2005-05; Primary Completion 2008-05 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Bronchopulmonary dysplasia | 36 weeks of life

CONTACTS AND LOCATIONS:
Overall Officials: Michele C. Walsh, MD MS, Principal Investigator — Case Western Reserve University, Rainbow Babies & Children's Hospital; Abbot R. Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Kurt Schibler, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Ronald N. Goldberg, MD, Principal Investigator — Duke University; Barbara J. Stoll, MD, Principal Investigator — Emory University; Brenda B. Poindexter, MD MS, Principal Investigator — Indiana University; Krisa P. Van Meurs, MD, Principal Investigator — Stanford University; Ivan D. Franz, III, MD, Principal Investigator — Tufts Medical Center; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Neil N. Finer, MD, Principal Investigator — University of California, San Diego; Edward F. Bell, MD, Principal Investigator — University of Iowa; Charles R. Bauer, MD, Principal Investigator — University of Miami; Kristi L. Watterberg, MD, Principal Investigator — University of New Mexico; Dale L. Phelps, MD, Principal Investigator — University of Rochester; Roger G. Faix, MD, Principal Investigator — University of Utah; Pablo J. Sanchez, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Kathleen A. Kennedy, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; T. Michael O'Shea, MD MPH, Principal Investigator — Wake Forest University; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; Abhik Das, PhD, Principal Investigator — RTI International
Locations (21):
- United States (21):
  - University of Alabama, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - University of California at San Diego, San Diego, California
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - Wake Forest University, Charlotte, North Carolina
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Walsh MC, Yao Q, Gettner P, Hale E, Collins M, Hensman A, Everette R, Peters N, Miller N, Muran G, Auten K, Newman N, Rowan G, Grisby C, Arnell K, Miller L, Ball B, McDavid G; National Institute of Child Health and Human Development Neonatal Research Network. Impact of a physiologic definition on bronchopulmonary dysplasia rates. Pediatrics. 2004 Nov;114(5):1305-11. doi: 10.1542/peds.2004-0204. PMID 15520112
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/